CLINICAL TRIAL: NCT00445939
Title: A Multi-Center, Randomized, Double-blind, Placebo-controlled Study of Adalimumab for the Induction of Clinical Remission in Japanese Subjects With Crohn's Disease
Brief Title: A Study of Adalimumab for the Induction of Clinical Remission in Japanese Subjects With Crohn's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M04-729
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2009-03-23 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Adalimumab 160 mg/80 mg (Experimental)
  Interventions: Biological: adalimumab
- Adalimumab 80 mg/40 mg (Experimental)
  Interventions: Biological: adalimumab
- Placebo (Placebo Comparator)
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: adalimumab — 160 mg at Week 0, 80 mg at Week 2
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 160 mg/80 mg
Biological: adalimumab — 80 mg at Week 0, 40 mg at Week 2
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 80 mg/40 mg
Biological: placebo — Placebo at Week 0 and Week 2
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of adalimumab for the induction of clinical remission in Japanese subjects with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's Disease Activity Index (CDAI) score of >= 220 and <= 450
* If subjects have previously been administered infliximab, subjects who discontinued use due to a loss of response or intolerance to infliximab therapy

Exclusion Criteria:

* Ulcerative colitis or indeterminate colitis
* History of cancer, lymphoma, leukemia or lymphoproliferative disease, active tuberculosis (TB), or Human immunodeficiency virus (HIV)
* Body weight is below 30 kg
* Surgical bowel resections within the past 6 months
* Females who are pregnant or breast-feeding or considering becoming pregnant during the study

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morio Ozawa, Study Director — Abbott Japan Co.,Ltd
Locations (18):
- Japan (18):
  - Aichi
  - Chiba
  - Ehime
  - Fukuoka
  - Hiroshima
  - Hokkaido
  - Hyōgo
  - Kagawa
  - Kanagawa
  - Kochi
  - Kyoto
  - Miyagi
  - Okayama
  - Okinawa
  - Osaka
  - Shiga
  - Shizuoka
  - Tokyo

REFERENCES:
- [Derived] Watanabe M, Hibi T, Lomax KG, Paulson SK, Chao J, Alam MS, Camez A; Study Investigators. Adalimumab for the induction and maintenance of clinical remission in Japanese patients with Crohn's disease. J Crohns Colitis. 2012 Mar;6(2):160-73. doi: 10.1016/j.crohns.2011.07.013. Epub 2011 Aug 26. PMID 22325170

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with moderate to severe Crohn's Disease (Crohn's Disease Activity Index [CDAI] >= 220 and <= 450) were enrolled into study. The period from the first dose of study drug to the evaluation at Week 4 is Period A. The period from the study drug injection at Week 4 to the evaluation at Week 8 is Period B.
Pre-assignment Details: All subjects were evaluated at Week 4. If responders (CDAI decrease >= 70 points compared to Baseline), rolled over to a maintenance study. If non-responders (CDAI decrease of < 70 points compared to Baseline), continued in study and received: adalimumab 160/80 mg + 40/40 mg, or adalimumab 80/40 mg + 40/40 mg or placebo + adalimumab 160/80 mg.
Groups:
- Adalimumab 160 mg/80 mg: Adalimumab 160 mg at Week 0, 80 mg at Week 2
- Adalimumab 80 mg/40 mg: Adalimumab 80 mg at Week 0, 40 mg at Week 2
- Placebo: Placebo at Week 0, placebo at Week 2
- Adalimumab 40mg /40 mg: Non-responders continued after 4 weeks, Adalimumab 160 at Week 0, 80 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6; Adalimumab 80 mg at Week 0, 40 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6.
Period: Period A - Week 0 - Week 4
Arm/Group | Adalimumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Adalimumab 40mg /40 mg
Started | 33 | 34 | 23 | 0
Completed | 32 (23 rated as responders and 9 rated as non-responders in evaluation on Week 4.) | 32 (20 rated as responders and 12 rated as non-responders in evaluation on Week 4.) | 23 (7 rated as responders and 16 rated as non-responders in evaluation on Week 4.) | 0
Not Completed | 1 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Period: Period B - Week 4 - Week 8
Arm/Group | Adalimumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Adalimumab 40mg /40 mg
Started | 16 (Non-responders continued after 4 weeks, previous 16 placebo subjects allocated to 160/80 mg group.) | 0 (Non-responders continued after 4 weeks, previous 80/40 mg subjects allocated to 40/40 mg group.) | 0 (Non-responders continued after 4 weeks, previous placebo subjects allocated to 160/80 mg group.) | 21 (Non-responders continued after 4 weeks, previous 160/80 and 80/40 subjects allocated to 40/40 group.)
Completed | 14 | 0 | 0 | 20
Not Completed | 2 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo at Week 0, placebo Week 2
- Total: Total of all reporting groups
Arm/Group | Adalimumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Total
Number analyzed (Participants) | 33 | 34 | 23 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.60) | 30.6 (9.26) | 30.4 (6.93) | 31.1 (8.80)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender, Male/Female who received first dose of study drug
  Participants
    Female | 13 | 18 | 7 | 38
    Male | 20 | 16 | 16 | 52
Region of Enrollment [Number; unit: participants]
  Japan | 33 | 34 | 23 | 90

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With a Clinical Remission (Crohn's Disease Activity Index [CDAI] < 150) at Week 4
Description: CDAI is used to quantify the symptoms of patients with Crohn's Disease. A score below 150 indicates remission and a score above 450 indicates severe disease. Comparison of the number of subjects with a clinical remission (CDAI < 150) in the adalimumab 160 mg (Week 0)/ 80 mg (Week 2) and adalimumab 80 mg (Week 0)/ 40 mg (Week 2) groups at Week 4.
Time Frame: 4 Weeks
Population: The primary analysis will be performed on the full analysis set (randomized subjects who received at least one dose of study drug) using the non-responder imputation for missing remission observations.
Measure: Number; unit: Particpants
Arm/Group | Adalimumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo
Number analyzed (Participants) | 33 | 34 | 23
Particpants | 11 | 6 | 3

2. Secondary Outcome: Clinical Remission (CDAI < 150) at Week 2
Description: Number of subjects in each treatment group in clinical remission (CDAI < 150) in Full Analysis Set (FAS) using non-responder Imputation (NRI) at Week 2.
Time Frame: Week 2
Population: Subjects with a clinical remission (CDAI <= 150) in the adalimumab 160 mg (Week 0/80 mg (Week 2) and adalimumab 80 mg (Week 0)/40 mg (Week 2) in full analysis set using Non-responder Imputation.
Measure: Number; unit: Participants
Groups:
- Adaliumab 160 mg/80 mg: Adalimumab 160 mg at Week 0, 80 mg at Week 2
- Placebo + 160/80 mg: Placebo at Week 0, placebo at Week 2
Arm/Group | Adaliumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo + 160/80 mg
Number analyzed (Participants) | 33 | 34 | 23
Participants
  Week 2 | 6 | 5 | 1

3. Secondary Outcome: Clinical Response (CR-70 and CR-100) in Period A
Description: The number of subjects in each treatment group with a clinical response 70 (CDAI decrease of >=70 compared to Baseline) and 100 (CDAI decrease of >=100 compared to Baseline) at Week 2 and Week 4.
Time Frame: Weeks 2 and Week 4
Population: The secondary efficacy analysis was performed using descriptive statistics in randomized subjects who received at least one dose of study drug (full analysis set) in the three treatment groups: Adalimumab 160 mg/80 mg, adalimumab 80mg/40 mg, and placebo.
Measure: Number; unit: participants
Groups:
- Placebo: Placebo at Week 0, placebo at Week 2,
Arm/Group | Adaliumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo
Number analyzed (Participants) | 33 | 34 | 23
participants
  CR-70 at Week 2 | 15 | 17 | 4
  CR-70 at Week 4 | 23 | 20 | 7
  CR-100 at Week 2 | 10 | 11 | 2
  CR-100 at Week 4 | 15 | 17 | 4

4. Secondary Outcome: Clinical Response (CR-70 and CR-100) in Period B
Description: The Number of subjects in each treatment group with a CR-70 (CDAI decrease of >= 70 compared to Baseline) and 100 (CDAI decrease of >= 100 compared to Baseline) in subjects who were non-responders at Week 4 at Week 6 and Week 8.
Time Frame: Week 6 and Week 8
Population: Full analysis set - subjects rated as non-responders (did not attain CDAI reduction >= 70) in the evaluation of CR-70 and CR-100 at Week 4. For Week 6 and Week 8 descriptive statistics performed only for non-responders at Week 4 in the three treatment groups: adalimumab 160/80 mg + 40/40 mg, adalimumab 80/40 mg + 40/40 mg, and placebo + 160/80 mg.
Measure: Number; unit: Participants
Groups:
- Adaliumab 160 mg/80 mg + 40/40 mg: Adalimumab 160 mg at Week 0, 80 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6
- Adalimumab 80 mg/40 mg + 40/40 mg: Adalimumab 80 mg at Week 0, 40 mg at Week 2, 40 mg at Week 4, and 40 mg at Week 6
- Placebo + Adalimumab 160/80 mg: Placebo at Week 0, placebo at Week 2, adalimumab 160 mg at Week 4, and adalimumab 80 mg at Week 6
Arm/Group | Adaliumab 160 mg/80 mg + 40/40 mg | Adalimumab 80 mg/40 mg + 40/40 mg | Placebo + Adalimumab 160/80 mg
Number analyzed (Participants) | 9 | 12 | 16
Participants
  CR-70 at Week 6 | 1 | 4 | 9
  CR-70 at Week 8 | 3 | 5 | 12
  CR-100 at Week 6 | 0 | 1 | 3
  CR-100 at Week 8 | 0 | 2 | 7

5. Secondary Outcome: Clinical Remission (CDAI <150) at Week 6 and Week 8
Description: The number of subjects with clinical remission (CDAI < 150) in the subjects who were non-responders at Week 4 calculated with non-responder imputation (NRI) at Week 6 and Week 8
Time Frame: Week 6 and Week 8
Population: Subjects who were rated as non-responders (CDAI reduction < 70) in the evaluation of clinical remission (CDAI<150) at Week 4. For Week 6 and Week 8 descriptive statistics performed only for non-responders at Week 4 in the three treatment groups: adalimumab 160/80 mg + 40/40 mg, adalimumab 80/40 mg + 40/40 mg, and placebo + adalimumab 160/80 mg.
Measure: Number; unit: Participants
Groups:
- Adaliumab 160 mg/80 mg + 40/40 mg: Adalimumab 160 mg at Week 0, 80 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6
- Adalimumab 80 mg/40 mg + 40/40 mg: Adalimumab 80 mg at Week 0, 40 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6
- Placebo + Adalimumab 160/80 mg: Placebo at Week 0, placebo at Week 2, 160 mg at Week 4, 80 mg at Week 6
Arm/Group | Adaliumab 160 mg/80 mg + 40/40 mg | Adalimumab 80 mg/40 mg + 40/40 mg | Placebo + Adalimumab 160/80 mg
Number analyzed (Participants) | 33 | 34 | 23
Participants
  Clinical Remission at Week 6 | 0 | 1 | 2
  Clinical Remission at Week 8 | 0 | 1 | 2

ADVERSE EVENTS:
Groups:
- Adalimumab 160 mg/80 mg + 40/40 mg: Adalimumab 160 mg at Week 0, 80 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6
- 80/40 mg + 40/40 mg: Adalimumab 80 mg at Week 0, 40 mg at Week 2, 40 mg at Week 4, 40 mg at Week 6
Arm/Group | Adaliumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Adalimumab 160 mg/80 mg + 40/40 mg | 80/40 mg + 40/40 mg | Placebo + Adalimumab 160/80 mg
Serious Adverse Events (participants affected / at risk) | 1 | 3 | 2 | 1 | 1 | 0
Other Adverse Events (participants affected / at risk) | 12 | 15 | 8 | 5 | 9 | 8
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Adaliumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Adalimumab 160 mg/80 mg + 40/40 mg | 80/40 mg + 40/40 mg | Placebo + Adalimumab 160/80 mg
Abdominal abcess (Infections and infestations) | 0/33 | 1/34 | 0/23 | 0/9 | 0/12 | 0/16
C-reactive protein increased (at investigator's discretion) (Investigations) | 0/33 | 1/34 | 0/23 | 0/9 | 0/12 | 0/16
Crohn's Disease (Gastrointestinal disorders) | 0/33 | 2/34 | 2/23 | 1/9 | 1/12 | 0/16
Epididymitis (Reproductive system and breast disorders) | 1/33 | 0/34 | 0/23 | 0/9 | 0/12 | 0/16
Subileus (Gastrointestinal disorders) | 0/33 | 1/34 | 0/23 | 0/9 | 0/12 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Adaliumab 160 mg/80 mg | Adalimumab 80 mg/40 mg | Placebo | Adalimumab 160 mg/80 mg + 40/40 mg | 80/40 mg + 40/40 mg | Placebo + Adalimumab 160/80 mg
Abdominal distension (Gastrointestinal disorders) | 2/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Abdominal pain (Gastrointestinal disorders) | 0/33 | 0/34 | 1/23 | 0/9 | 1/12 | 0/16
Adverse drug reaction (General disorders) | 1/33 | 1/34 | 1/23 | 1/9 | 0/12 | 0/16
Alopecia (Skin and subcutaneous tissue disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Anaemia (Blood and lymphatic system disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Antinuclear antibody increased (at investigator's discretion) (Investigations) | 0/33 | 1/34 | 0/23 | 0/9 | 1/12 | 0/16
Application site swelling (General disorders) | 0/33 | 0/34 | 0/23 | 1/9 | 0/12 | 0/16
Back pain (Musculoskeletal and connective tissue disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Blood albumin decreased (at investigator's discretion) (Investigations) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Blood creatine phosphokinase (at investigator's discretion) (Investigations) | 0/33 | 1/34 | 0/23 | 1/9 | 0/12 | 0/16
Blood glucose increased (at investigator's discretion) (Investigations) | 2/33 | 0/34 | 0/23 | 0/9 | 0/12 | 0/16
Chest pain (General disorders) | 0/33 | 0/34 | 0/23 | 1/9 | 0/12 | 0/16
Constipation (Gastrointestinal disorders) | 2/33 | 0/34 | 1/23 | 0/9 | 0/12 | 0/16
Diarrhoea (Gastrointestinal disorders) | 0/33 | 0/34 | 1/23 | 0/9 | 1/12 | 0/16
Dry skin (Skin and subcutaneous tissue disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Feeling abnormal (General disorders) | 0/33 | 0/34 | 0/23 | 1/9 | 0/12 | 0/16
Glucose tolerance impaired (at investigator's discretion) (Metabolism and nutrition disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Haemorrhoids (Gastrointestinal disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Headache (Nervous system disorders) | 3/33 | 0/34 | 1/23 | 0/9 | 2/12 | 1/16
Hepatic function abnormal (Hepatobiliary disorders) | 1/33 | 2/34 | 0/23 | 0/9 | 0/12 | 0/16
Herpes Simplex (Infections and infestations) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Hypersensitivity (Immune system disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Hypoglycaemia (Metabolism and nutrition disorders) | 0/33 | 0/34 | 0/23 | 1/9 | 0/12 | 0/16
Injection site erythema (General disorders) | 2/33 | 0/34 | 0/23 | 0/9 | 0/12 | 0/16
Injection site pain (General disorders) | 1/33 | 2/34 | 0/23 | 0/9 | 0/12 | 0/16
Injection site reaction (General disorders) | 1/33 | 3/34 | 2/23 | 0/9 | 1/12 | 0/16
Instillation site pain (General disorders) | 0/33 | 0/34 | 0/23 | 1/9 | 0/12 | 0/16
Intestinal obstruction (Gastrointestinal disorders) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0/33 | 1/34 | 0/23 | 1/9 | 0/12 | 1/16
Malaise (General disorders) | 0/33 | 3/34 | 0/23 | 0/9 | 0/12 | 0/16
Nasopharyngitis (Infections and infestations) | 0/33 | 1/34 | 0/23 | 1/9 | 1/12 | 3/16
Nausea (Gastrointestinal disorders) | 1/33 | 1/34 | 3/23 | 0/9 | 0/12 | 0/16
Pyrexia (General disorders) | 1/33 | 2/34 | 0/23 | 0/9 | 0/12 | 0/16
Rash (Skin and subcutaneous tissue disorders) | 2/33 | 0/34 | 1/23 | 0/9 | 0/12 | 0/16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0/33 | 3/34 | 0/23 | 0/9 | 0/12 | 0/16
Thermal burn (Injury, poisoning and procedural complications) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Tonsillitis (Infections and infestations) | 0/33 | 0/34 | 0/23 | 0/9 | 1/12 | 0/16
Upper respiratory tract infection (Infections and infestations) | 3/33 | 1/34 | 1/23 | 1/9 | 0/12 | 0/16
Urinary tract infection (Infections and infestations) | 0/33 | 0/34 | 0/23 | 0/9 | 0/12 | 1/16
Vomiting (Gastrointestinal disorders) | 2/33 | 0/34 | 1/23 | 0/9 | 0/12 | 0/16

LIMITATIONS AND CAVEATS:
Small population, therefore no statistical tests were performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; most restrictive agreement states Medical Institution shall not disclose materials/information disclosed by Abbott Japan in connection with the Clinical Research, or information obtained by conducting the Clinical Research, to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting the Clinical Research, Medical Institution shall obtain Abbott Japan's prior written approval.